CLINICAL TRIAL: NCT01839539
Title: Phase Ⅱ Study of Dendritic and Cytokine-induced Killer Cells (DC-CIK) Treatment in Patients With Stage Ⅲ Colorectal Cancer
Brief Title: Study of DC-CIK to Treat Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Weiliang Sun, Investigator, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRC-01
Record Dates: First submitted 2013-04-14; First posted 2013-04-25 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; DC-CIK; CRC
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (No Intervention): After neoadjuvant and (or) adjuvant chemotherapy or (and) radiotherapy according to NCCN guidelines, patients will only regularly follow up.
- A (Experimental): After neoadjuvant and (or) adjuvant chemotherapy or (and) radiotherapy according to NCCN guidelines, patients will receive 2-3 cycles of Dendritic and Cytokine-induced Killer Cells (DC-CIK) treatment (every 4 weeks).
  Interventions: Biological: dendritic and cytokine-induced killer cells

INTERVENTIONS:
Biological: dendritic and cytokine-induced killer cells
  Other Names: DC-CIK
  Arms: A

SUMMARY:
The purpose of this study is to evaluate the efficacy of dendritic and cytokine-induced killer cells (DC-CIK) for colorectal cancer (CRC).

DETAILED DESCRIPTION:
60 patients with stage Ⅲ CRC, who had received neoadjuvant and (or) adjuvant chemotherapy or (and) radiotherapy according to NCCN guidelines, and got complete response (CR), will be randomly divided into group A (receive DC-CIK treatment) or group B (just regularly follow up), and the randomize ratio will be 1:1. Patients in group A will receive 2-3 cycles of DC-CIK cells treatment (every 4 weeks). Patients in group B will have no anti-tumor therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age;
2. CRC with histological diagnose, and had received neoadjuvant and (or) adjuvant chemotherapy or (and) radiotherapy and got complete response (CR) with imaging;
3. Patients who have a life expectancy of at least 3 months;
4. Eastern Cooperative Oncology Group (ECOG) performance status was 0 - 1;
5. The bone marrow functioned normally (WBC > 4.0×109/L, Hb > 120 g/L, PLT > 100×109/L);
6. The ECG results were normal, and the liver and kidney were functional.

Exclusion Criteria:

1. Patients who had distant metastases;
2. Patients with uncontrolled infection; underlying disease that was severe or life-threatening;
3. Patients who were pregnant or lactating;
4. ECOG perform status ≥ 2;
5. Patients who are suffering from auto immune diseases or patients who need to accept glucocorticoid treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 5 years

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
Quality of life (QOL) | 5 years
Laboratory findings (The number of CD3+ (or CD8+ or CD4+ or CD56+)T cell) | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Guangxi Medical University, Nanning, Guangxi, China